CLINICAL TRIAL: NCT05726994
Title: Volatilomic Approaches for the Study of CFTR Modulators
Brief Title: Volatilomic Approaches for the Study of CFTR Modulators (VOLATIL-CF)
Acronym: VOLATIL-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221173
Record Dates: First submitted 2023-01-12; First posted 2023-02-14 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; volatile organic compounds (VOC); exhaled breath; CFTR modulators
MeSH Terms: conditions — Cystic Fibrosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced sputum, Plasma, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cystic fibrosis and Kaftrio®: 20 children with cystic fibrosis aged 6 to 12 who initiate Kaftrio®
  Interventions: Biological: exhaled breath collection; Other: Data collection

INTERVENTIONS:
Biological: exhaled breath collection — Fasting children will be asked to breathe normally through a mouthpiece for the collection and analysis of exhaled breath.
Other: Data collection — Clinical data will be collected in order to seek correlations with the exhaled breath profile.

SUMMARY:
This study relies on the hypotheses that (1) exhaled breath is intimately correlated to the patient's lung condition and that (2)the composition of exhaled breath , i.e. the VOCs profile, will be significantly modified from the first days of treatment by CFTR modulators in a or pauci/symptomatic patients such as young children under 12 years old. The non-invasive and longitudinal collection and analysis of exhaled breath may reveal modifications in signaling pathways impacted by these treatments on the very short term. This study is a single-center pilot study.

DETAILED DESCRIPTION:
This is a single-center prospective cohort study that plans to include 20 children with cystic fibrosis aged 6 to 12 years old who will initiate Kaftrio® in early 2023.

The children will be monitored for one month; three visits are planned as part of routine care (before initiation of treatment, in the course of the first week and after one month of treatment) during which exhaled breath collection and analysis will also be performed. Access to clinical data collected throughout routine follow-up of these children (analysis of induced sputum, urine and blood, sweat test, respiratory function tests) will be granted upon patient/parent authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis initiating Kaftrio® treatment.
* Patients and holders of parental authority not opposing participation in this research.
* Patients affiliated to a Health Insurance system or beneficiaries. Exclusion Criteria
* Patients deprived of liberty or under guardianship.
* Pregnant or breastfeeding patients.
* Lung transplanted patients.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Children with cystic fibrosis aged 6 to 12 who will start Kaftrio® treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
volatile organic compounds (VOC) profile | At 0 day, 7 days, and 1 month of treatment
  identification of VOCs in exhaled breath with a significant variation between 0 day, 7 days, and/or 1 month of treatment

SECONDARY OUTCOMES:
Weight | At 0 day, 7 days, and 1 month of treatment
  Weight measured at visits
Sweat test | At 0 day, 7 days, and 1 month of treatment
  Sweat test result
Induced sputum - microbiology | At 0 day, 7 days, and 1 month of treatment
  Results of microbiological analysis of induced sputum
Induced sputum - immunology | At 0 day, 7 days, and 1 month of treatment
  Results of inflammatory markers analysis of induced sputum (neutrophil elastase, IL-8, IL-1b, IL-6)
Spirometry | At 0 day, 7 days, and 1 month of treatment
  Results of spirometry FVC measurements
Spirometry | At 0 day, 7 days, and 1 month of treatment
  Results of spirometry FEV1 measurements
Spirometry | At 0 day, 7 days, and 1 month of treatment
  Results of spirometry DEM25-75 measurements
Urine | At 0 day and 1 month of treatment
  Biobanking for metabolic study
Blood | At 0 day and 1 month of treatment
  Biobanking for metabolic study

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle SERMET-GAUDELUS, Professor, Study Director — APHP
Locations (1):
- Hôpital Necker - Enfants malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No